CLINICAL TRIAL: NCT02830165
Title: Phase I Feasibility Trial of Preoperative Adjuvant Stereotactic Body Radiotherapy for Patients at High Risk of Local Failure After Prostatectomy
Brief Title: Stereotactic Body Radiation Therapy in Treating Patients With High-Risk Prostate Cancer Undergoing Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-001580; NCI-2016-00188 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); JCCCID608; P50CA092131 (NIH)
Record Dates: First submitted 2016-07-07; First posted 2016-07-12 (Estimated); Results first posted 2022-01-06 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2022-05

CONDITIONS: Stage I Prostate Adenocarcinoma American Joint Committee on Cancer (AJCC) v7; Stage II Prostate Adenocarcinoma AJCC v7; Stage III Prostate Adenocarcinoma AJCC v7
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (SBRT) (Experimental): Patients undergo 3 fractions of SBRT over 1-2 weeks, 2-4 weeks prior to radical prostatectomy.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This phase I trial studies stereotactic body radiation therapy (SBRT) in treating patients with prostate cancer that is likely to come back or spread (high-risk) undergoing surgery. Stereotactic body radiation therapy uses special equipment to position a patient and deliver radiation to tumors with high precision. This method can kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue. Delivering radiotherapy before prostatectomy by SBRT is more convenient, conformal, and may spare normal tissues better than delivering radiotherapy after prostatectomy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess feasibility of pre-operative stereotactic body radiotherapy (SBRT) in prostate cancer patients at high risk for recurrence after prostatectomy.

SECONDARY OBJECTIVES:

I. To assess safety and acute toxicity of SBRT followed by prostatectomy. This will be based on Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 and patient reported quality of life (Expanded Prostate Cancer Index Composite [EPIC] and International Prostate Symptom Score [IPSS] questionnaires).

II. Investigation of the radiobiology of SBRT in prostate cancer using resected prostate tumor tissue.

III. Evaluation of the nature of the immune response to prostate cancer generated by SBRT.

OUTLINE:

Patients undergo 3 fractions of SBRT over 1-2 weeks, 2-4 weeks prior to radical prostatectomy.

After completion of the study treatment, patients are followed up at 0 to 4 weeks, and every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary non-metastatic adenocarcinoma of the prostate
* Patient desires and is medically fit to undergo prostatectomy
* Karnofsky performance status (KPS) >= 70
* Patients on androgen deprivation therapy (ADT) are allowed
* For confirmation of high risk local failure status, patients will have any one of the following:

  * Computed tomography (CT) or magnetic resonance imaging (MRI) demonstrating seminal vesicle invasion (SVI) or extraprostatic extension (EPE) within 1 year of enrollment into the study
  * Pre-biopsy prostate-specific antigen (PSA) >= 20
  * Gleason score 7-10 (Gleason 7 must be 4+3), presence of any Gleason 5 (even if a tertiary score) as determined at diagnostic biopsy
  * Gleason score 7 and > 50% of biopsy cores positive for prostate cancer
  * Clinical stage >= T3 (staging by imaging acceptable)
* An image-guided biopsy (via Artemis Ultrasound with MRI co-registration) is encouraged but not required if not performed as standard of care biopsy

Exclusion Criteria:

* Distant metastases, based upon:

  * CT scan or MRI of the abdomen/pelvis or prostate specific membrane antigen (PSMA) positron emission tomography/computed tomography (PET/CT) within 120 days prior to registration and
  * Bone scan or PSMA PET/CT within 120 days prior to registration; if the bone scan is suspicious, a plain x-ray and/or MRI must be obtained to rule out metastasis prior to registration
* Patient is unable or unwilling to sign consent
* Patient is considered low-risk and would not have received adjuvant radiation therapy (RT) outside of this study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2020-05-09 (Actual); Study Completion 2022-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Nickols, MD, PhD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was open to recruitment from 6/15/2016 and closed to enrollment 09/08/2019
Groups:
- Stereotactic Body Radiation Therapy (SBRT): Patients undergo 3 fractions of stereotactic body radiation therapy (SBRT) over 1-2 weeks, 2-4 weeks prior to radical prostatectomy.
Period: Overall Study
Arm/Group | Stereotactic Body Radiation Therapy (SBRT)
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Stereotactic Body Radiation Therapy (SBRT): Patients undergo 3 fractions of SBRT over 1-2 weeks, 2-4 weeks prior to radical prostatectomy.
Arm/Group | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11
Gleason Grade [Count of Participants; unit: Participants] — Gleason grade assigned based on predominant pattern in biopsy + a second Gleason grade to the second most predominate pattern. The two grades are added together to determine the Gleason score. Assigned Gleason scores range from 6 - 10, with 6 being low grade or better and 10 is high grade or worse.
  Participants
    Gleason 9 | 3
    Gleason 8 | 5
    Gleason 7 | 3
CStage [Count of Participants; unit: Participants] — Primary tumor, regional nodes, metastasis (TNM) staging system: A system to describe the amount and spread of cancer in a patient's body, using TNM. T describes the size of the tumor and any spread of cancer into nearby tissue; N describes spread of cancer to nearby lymph nodes; and M describes metastasis (spread of cancer to other parts of the body). Larger numbers indicate worse indication.
  Participants
    cT1cNoMo | 2
    cT1cN1Mo | 1
    cT2aNoMo | 2
    cT2bNoMo | 2
    cT2cN1Mo | 1
    cT3aNoMo | 1
    cT3aN1Mo | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed the Maximum Time Allowed on Study Without Severe Acute Surgical Complications
Time Frame: At 4 weeks post surgery
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Stereotactic Body Radiotherapy (SBRT): Patients undergo 3 fractions of SBRT over 1-2 weeks, 2-4 weeks prior to radical prostatectomy.
Arm/Group | Treatment Stereotactic Body Radiotherapy (SBRT)
Number analyzed (Participants) | 11
Participants | 11

2. Secondary Outcome: Number of Participants With Genitourinary Toxicities and Gastrointestinal Toxicities
Description: Based on the Common Terminology Criteria for Adverse Events (CTCAE) v4. Grade refers to the severity of the adverse event. Indications are Grade 1 is Mild, Grade 2 is Moderate, Grade 3 is Severe or medically significant but not immediately life threatening. Grade 0 refers to absence of an adverse event (ae).
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 11
Participants
  Genitourinary Toxicities: Grade 0 | 1
  Genitourinary Toxicities: Grade 1 | 4
  Genitourinary Toxicities: Grade 2 | 4
  Genitourinary Toxicities: Grade 3 | 2
  Gastrointestinal toxicities: Grade 0 | 9
  Gastrointestinal toxicities: Grade 1 | 1
  Gastrointestinal toxicities: Grade 2 | 1
  Gastrointestinal toxicities: Grade 3 | 0

3. Secondary Outcome: Changes in Quality of Life (QOL) ,From Baseline to 12 Months, as Measured on the Expanded Prostate Cancer Index Composite (EPIC-26) Questionnaire Scoring.
Description: The Expanded Prostate Cancer Index Composite Short Form (EPIC-26) is composed of 26 items and measures health-related quality of life across 5 prostate cancer domains. Response options for each EPIC item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing a better quality of life.
Time Frame: score from baseline to twelve months
Population: Mean change in EPIC-26 score from baseline to 12 months. Three patients dd not complete the QOL assessment and therefore were not included in the analysis.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Treatment Stereotactic Body Radiotherapy (SBRT): Change in score from baseline at 12 months. Quality-of-Life Assessment: Ancillary studies
Arm/Group | Treatment Stereotactic Body Radiotherapy (SBRT)
Number analyzed (Participants) | 8
score on a scale
  Urinary Incontinence | -32.8 [-55.3 to -10.3]
  urinary irritative/obstructive | -1.6 [-9.6 to 6.4]
  Bowel | -2.1 [-8.2 to 4]
  Sexual Function | -34.4 [-49.4 to -19.4]
  Hormonal | -10.6 [-26.0 to 4.8]

4. Secondary Outcome: Changes in Quality of Life as Measured on the International Prostate Symptom Score (IPSS) Questionnaire.
Description: The International Prostate Symptom Score is composed of seven questions and scored from 0 - 35, with higher scores indicating more severe symptoms.
Time Frame: Mean change in I-PSS score from baseline to 12 months.
Population: Three patients dd not complete the QOL assessment and therefore were not included in the analysis.
Measure: Mean (95% Confidence Interval); unit: change in score on a scale
Arm/Group | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 8
change in score on a scale | 0.5 [-2.1 to 3.1]

5. Secondary Outcome: Correlative Biomarker Analyses Using Tissue and Serial Blood Samples
Description: Tissue specimens of the primary tumor as well as blood draws before and after treatment will be used to conduct biomarker and molecular analyses relevant to understanding the biology of prostate SBRT
Time Frame: Baseline and to up to 1 year
Population: Pre-treatment biopsies and surgical specimens from this trial were used to determine radiation-induced changes in macrophage subsets. Six participants had available paired biopsy cores and Radical Prostatectomy (RP) specimens for analysis.
Measure: Mean (Standard Deviation); unit: Macropahge cells per pixel area
Groups:
- Post SBRT and Radical Prostatectomy (RP): Patients undergo 3 fractions of SBRT over 1-2 weeks, 2-4 weeks prior to radical prostatectomy.
Arm/Group | Stereotactic Body Radiation Therapy (SBRT) | Post SBRT and Radical Prostatectomy (RP)
Number analyzed (Participants) | 6 | 6
Macropahge cells per pixel area
  CD11b | 0.002 (.07) | 0.004 (.01)
  CD68 | 0.01 (.05) | 0.035 (.01)
  CD163 | 0.005 (.05) | 0.03 (.07)

6. Secondary Outcome: Correlative Biomarker Analyses Using Tissue and Serial Blood Samples
Description: as for outcome 5
Time Frame: Baseline and to up to 1 year
Population: Pre-treatment biopsies and surgical specimens from this trial were used to determine radiation-induced changes in T cell. Six participants had available paired biopsy cores and RP specimens for analysis.
Measure: Mean (Standard Deviation); unit: cells per Tumor area mm2
Arm/Group | Stereotactic Body Radiation Therapy (SBRT) | Post SBRT and Radical Prostatectomy (RP)
Number analyzed (Participants) | 6 | 6
cells per Tumor area mm2
  CD3+CD8 | 70 (15) | 30 (10)
  CD3+CD4 | 110 (10) | 90 (20)
  CD4+FOXp3 | 30 (10) | 50 (15)

ADVERSE EVENTS:
Time Frame: 90 day intervals for 1 year
Arm/Group | Stereotactic Body Radiation Therapy (SBRT)
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 2/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stereotactic Body Radiation Therapy (SBRT) (N=11)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stereotactic Body Radiation Therapy (SBRT) (N=11)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Difficulty Urinating (Renal and urinary disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Erectile Dysfunction (General disorders) | 4 (4)
Hemorrhoids (Gastrointestinal disorders) | 2 (2)
Incontinence (Renal and urinary disorders) | 1 (1)
Increased Bowel Movement (Gastrointestinal disorders) | 1 (1)
Loose Bowel Movement (Gastrointestinal disorders) | 1 (1)
Loose Stools (Gastrointestinal disorders) | 1 (1)
Loss of Sexual Function (General disorders) | 1 (1)
Mild Pain (General disorders) | 1 (1)
Nocturia (Renal and urinary disorders) | 3 (3)
Painless Hematuria (General disorders) | 1 (1)
Radiation Colopathy and Proctopathy (General disorders) | 1 (1)
Rectal Bleeding (General disorders) | 1 (1)
Slight Burning when Urinating (General disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 7 (7)
Urinary Incontinence (Renal and urinary disorders) | 6 (8)
Urinary Tract Pain (Renal and urinary disorders) | 1 (1)
Urinary Urgency (Renal and urinary disorders) | 3 (3)
Abdominal Pain (General disorders) | 1 (1)
Anxiety (General disorders) | 2 (2)
Atrial Fibrillation (General disorders) | 1 (1)
Benign Polyp (General disorders) | 1 (1)
Bilateral Eye Irritation and Redness (Eye disorders) | 1 (1)
Chills (General disorders) | 2 (2)
Dyspenea (General disorders) | 1 (1)
Edema Suprepubic (General disorders) | 1 (1)
Fatigue (General disorders) | 5 (5)
Hot Flashes (General disorders) | 1 (1)
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lower Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Middle Mediastinal Schwannoma (General disorders) | 1 (1)
Muscle Aches (neck and shoulders) (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Perineal Numbness (General disorders) | 1 (1)
Pseudogout (Musculoskeletal and connective tissue disorders) | 1 (1)
Sweating (General disorders) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT02830165/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/65/NCT02830165/ICF_001.pdf